CLINICAL TRIAL: NCT01446744
Title: Stereotactic Ablative Radiotherapy for Comprehensive Treatment of Oligometastatic Tumors (SABR-COMET): A Randomized Phase II Trial
Brief Title: Stereotactic Ablative Radiotherapy for Comprehensive Treatment of Oligometastatic Tumors (SABR-COMET)
Acronym: SABR-COMET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Regional Cancer Program, Canada (Other); VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-11-605; SABR-COMET (Other: OCREB)
Record Dates: First submitted 2011-09-29; First posted 2011-10-05 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard arm (Active Comparator): Standard of care, palliative radiotherapy, and chemotherapy at the discretion of the treating medical oncologist
  Interventions: Radiation: palliative radiotherapy
- Stereotactic arm (Experimental): Stereotactic ablative radiotherapy, and chemotherapy at the discretion of the treating medical oncologist
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — Total dose and number of fractions will depend on the site of disease. Treatment will be given daily, or every other day, over 1 -3 weeks.
  Arms: Stereotactic arm
Radiation: palliative radiotherapy — Investigators should follow the principles of palliative radiotherapy as per the individual institution. Treatment recommendations are as follows:
  Brain: Whole brain radiotherapy i.e. 20 Gy in 5 fractions, 30 Gy in 10 fractions
  Lung: Palliative radiotherapy as per 2011 consensus guidelines.15 i.e. 8 Gy in 1 fraction, 20 Gy in 5 fractions, 30 Gy in 10 fractions
  Bone: Palliative radiotherapy as per 2011 consensus guidelines.16 i.e. 8 Gy in 1 fraction (most common), 20 Gy in 5 fractions, 30 Gy in 10 fractions
  Liver: 20 Gy in 5 fractions if standard institutional practice
  Arms: Standard arm

SUMMARY:
Stereotactic Ablative Radiotherapy (SABR) is a new radiation treatment that delivers high-dose, precise radiation to small tumors in 1-3 weeks of treatment. This new technique can potentially allow radiation treatments to be focused more precisely, and delivered more accurately than with older treatments. This improvement could help by reducing side effects and by improving the chance of controlling the cancer by more precisely treating the cancer. The purpose of this study is to compare SABR with current approaches of chemotherapy and conventional radiotherapy to assess the impact on overall survival and quality of life.

DETAILED DESCRIPTION:
TREATMENT PLAN

6.0.1 Standard Arm (Arm 1)

Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications. Patients in this arm should not receive stereotactic doses or radiotherapy boosts.

Treatment recommendations are as follows:

Brain: Whole brain radiotherapy i.e. 20 Gy in 5 fractions, 30 Gy in 10 fractions

Lung: Palliative radiotherapy as per 2011 consensus guidelines.15 i.e. 8 Gy in 1 fraction, 20 Gy in 5 fractions, 30 Gy in 10 fractions

Bone: Palliative radiotherapy as per 2011 consensus guidelines.16 i.e. 8 Gy in 1 fraction (most common), 20 Gy in 5 fractions, 30 Gy in 10 fractions

Liver: 20 Gy in 5 fractions if standard institutional practice

6.0.2 Treatment Planning for Standard Arm

Treatment planning is to be done using CT simulation or conventional simulation (fluoroscopy) as per individual institutional practice. Simple beam arrangements, such as parallel opposed beams, are favored wherever possible.

6.1 Experimental Arm (Arm 2)

All treatments in this study are based on current protocols in clinical use at the LRCP and VUmc for treatment of lung,17 liver,18 brain,19,20 and spinal cord21 metastases. The guiding principle for radiotherapy is to achieve disease control but to minimize any potential adverse impact on quality of life. Concurrent chemotherapy or targeted therapy at the time of radiotherapy is not permitted within the 4 weeks prior to SABR. Hormone therapy is permitted.

6.1.1 Dose/Fractionation

Lung- tumors 3 cm or less surrounded by lung parenchyma, 54(Gy) in 3 fractions

* Abutting chest wall or >3 cm, 55(Gy)in 5 fractions, every second day
* Within 2 cm of mediastinum or brachial plexus, 60(Gy),8* fractions, every second day

Bone -Any bone except femur,35(Gy), in 5 fractions,daily

* vertebral body,16-20(Gy)in 1 fraction, single dose, or 30Gy in 3 fractions, every second day

Brain - Non-radiosurgical,40(Gy) to metastases, in 5 fractions,daily

* If whole brain treated, then simultaneous boost to each lesion,20 Gy whole brain (optional), in 5 fractions, daily
* Radiosurgical, ≤1 cm, 22-24(Gy), in 1 fraction, >1 and ≤2 cm, 22-24(Gy) in 1 fraction >2 and ≤ 3 cm, 18-20(Gy) in 1 fraction Optional whole brain to follow (see text) Liver-LRCP site: Dose is based on calculated normal tissue probability of <5%,Every second day
* other sites 45-60(Gy), in 3-8 fractions, every second day

Adrenal, 60 (Gy), in 8 fractions, every second day

(If whole brain treated, then simultaneous boost to each lesion)

6.1.2 Immobilization

Treatment will be setup using reproducible positioning, verified using an on-line protocol, for all patients in this study. Immobilization may include a custom immobilization device, such as thermoplastic shell or vac-lok bag, as per individual institutional practice when delivering SABR. Some centers do not use immobilization devices and have demonstrated high degrees of accuracy; this is acceptable in this study.

6.1.3 Imaging/Localization/Registration All patients in Arm 2 will undergo planning CT simulation. 4-dimensional CT will be used for tumors in the lungs or liver. Axial CT images will be obtained throughout the region of interest. For centres using stereotactic radiosurgery platforms, real-time tumor tracking and orthogonal imaging systems are permitted.

Any center which is not yet experienced in lesions at any specific sub-site (e.g. adrenal metastases) shall be eligible to participate by including only patients with lesions at other pre-specified sites

It is strongly recommended that the doses to organs at risk are not to be exceeded - in some specific cases, this may require lower doses or higher fractionations than listed here. Such changes in dose will require approval of one of the local principal investigators. (see section 6.2)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* ECOG performance status 0-1
* Controlled primary tumor

  a. defined as: at least 3 months since original tumor treated definitively, with no progression at primary site
* All sites of disease can be safely treated based on criteria below
* Maximum 3 metastases in any single organ system (i.e. lung, liver, brain, bone)
* Life expectancy >6 months
* Not a candidate for surgical resection at all sites: surgery to all sites not recommended by multidisciplinary team, or unfit or declining surgery
* Prior chemotherapy allowed but no systemic therapy 4 weeks prior to first fraction of radiotherapy, during radiotherapy, or for two weeks after last fraction
* Patients with metastases that have been previously treated (e.g. prior resection, Radiofrequency Ablation (RFA) or radiotherapy):

  a. If that previously treated metastasis is controlled on imaging, the patient is eligible for this study and that site does not need treatment

  a. If that previously treated metastasis is NOT controlled on imaging:
  1. If the previous treatment was surgery, the patient is eligible if that site can be treated by SABR
  2. If the previous treatment was radiotherapy or RFA, the patient is ineligible.
* Patient presented at multidisciplinary tumor board or quality-assurance rounds.

Exclusion Criteria:

* Serious medical comorbidities precluding radiotherapy
* Bone metastasis in a femoral bone
* Patients with 1-3 brain metastasis and no disease elsewhere (these patients should not be randomized but treated with stereotactic radiotherapy as per results of randomized trials)
* Prior radiotherapy to a site requiring treatment
* Complete response to first-line chemotherapy (i.e. no measurable target for SABR)
* Malignant pleural effusion
* Inability to treat all sites of active disease
* Clinical or radiologic evidence of spinal cord compression OR tumor within 3 mm of spinal cord on Magnetic Resonance Imaging (MRI).
* Dominant brain metastasis requiring surgical decompression
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-11; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | At approximately end of year 4 (study completion)

SECONDARY OUTCOMES:
Quality of life: Assessed with the Functional Assessment of Cancer Therapy: General (FACT-G) | At approximately end of year 2, and end of year 4 (study completion)
Toxicity: Assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (e.g. liver, lung, bone) | At approximately the end of years 1, 2, 3, and 4 (study completion)
Progression-free survival | At approximately end of year 2, and end of year 4 (study completion)
Lesional control rate | At approximately end of year 2, and end of year 4 (study completion)
Number of cycles of further chemotherapy/systemic therapy | At approximately end of year 2, and end of year 4 (study completion)

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, PhD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute; Suresh Senan, MRCPFRCR,PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (10):
- Alfred Health, William Burkland Radiotherapy Centre, Melbourne, Victoria, Australia
- Canada (7):
  - BC Cancer Agency, Vancouver, British Columbia
  - Atlantic Clinical Cancer Research , QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Ottawa Cancer Centre, Ottawa, Ontario
  - PEI Cancer Treatment Center, Charlottetown, Prince Edward Island
  - McGill University Health Centre Research Institute, Montreal, Quebec
- VU University Amsterdam (VUmc), Amsterdam, Netherlands
- The Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

REFERENCES:
- [Derived] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Derived] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Derived] Palma DA, Haasbeek CJ, Rodrigues GB, Dahele M, Lock M, Yaremko B, Olson R, Liu M, Panarotto J, Griffioen GH, Gaede S, Slotman B, Senan S. Stereotactic ablative radiotherapy for comprehensive treatment of oligometastatic tumors (SABR-COMET): study protocol for a randomized phase II trial. BMC Cancer. 2012 Jul 23;12:305. doi: 10.1186/1471-2407-12-305. PMID 22823994